CLINICAL TRIAL: NCT03406871
Title: Regorafenib and Nivolumab Simultaneous Combination Therapy for Advanced and Metastatic Solid Tumors: Phase I Clinical Trial
Brief Title: Regorafenib and Nivolumab Simultaneous Combination Therapy
Acronym: REGONIVO
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kohei Shitara (Other)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry); Bayer Yakuhin, Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Kohei Shitara, Assistant Chief of Gastrointestinal Oncology Division, National Cancer Center Hospital East
Organization: National Cancer Center Hospital East (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPOC 1603 study
Record Dates: First submitted 2018-01-12; First posted 2018-01-23 (Actual); Results first posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2024-12

CONDITIONS: Advanced and Metastatic Solid Tumor
Keywords: Regorafenib; Nivolumab; Phase I clinical trial
MeSH Terms: conditions — Neoplasm Metastasis | interventions — regorafenib; Nivolumab

STUDY DESIGN:
Masking Description: Dose-escalation cohort: A total of 3-6 patients per level, for a total of 9-18 patients(Anticipated), 14(Actual) Expansion cohort: Approximately 30 patients in total, 36(Actual)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Level 1 (Active Comparator): Regorafenib: Oral administration at a dose of 80 mg given once per day for 21 consecutive days, with a 1-week washout period.
  Nivolumab: Given once every 2 weeks at a dose of 3.0 mg/kg via an intravenous infusion.
  When it is deemed that there is no problem with safety at the doses described above, tolerability will be verified at the level-2 dosages described below.
  Interventions: Drug: Regorafenib; Drug: Nivolumab
- Level 2 (Active Comparator): Regorafenib: Oral administration at a dose of 120 mg/day for 21 consecutive days, with a 1-week washout period.
  Nivolumab: Given once every 2 weeks at a dose of 3.0 mg/kg.
  When it is deemed that there is no problem with safety at the doses described above, tolerability will be verified at the level-3 dosages described below.
  Interventions: Drug: Regorafenib; Drug: Nivolumab
- Level 3 (Active Comparator): Regorafenib: Oral administration at a dose of 160 mg/day for 21 consecutive days, with a 1-week washout period.
  Nivolumab: Given once every 2 weeks at a dose of 3.0 mg/kg.
  After starting the trial, three cases are registered at level 1, and temporary case registration is suspended until safety evaluation of the first course is completed in all cases. If there are cases in which evaluation of DLT can not be performed properly, such as being canceled due to reasons other than safety during the course of the first course, the necessary number of cases is appropriately added to the administration level.
  Interventions: Drug: Regorafenib; Drug: Nivolumab
- Expansion cohort (Active Comparator): After completion of the final DLT evaluation period of the subjects in the dose escalating cohort, the decision to move the subjects into the expansion cohort will be determined once it is decided, upon deliberation between the sponsor and the principal investigator, that there are no problems associated with moving on. Furthermore, the opinion of the Data and Safety Monitoring Committee (DSMC) can be sought as required .
  Regarding the review of RD in the expansion cohort, please refer to "Analysis Population Description" in Primary Outcome Measures.
  Interventions: Drug: Regorafenib; Drug: Nivolumab

INTERVENTIONS:
Drug: Regorafenib — One course will last 28 days. Oral administration for 21 consecutive days, with a 1-week washout period. As for the expansion cohort, implemented using the RD estimated in the dose-escalation cohort.
  Other Names: Identification code of the investigational drug; BAY73-4506
Drug: Nivolumab — One course will last 28 days. Given once every 2 weeks at a dose of 3.0 mg/kg.
  Other Names: Identification code of the investigational drug; BMS-936558, MDX1106, ONO-4538

SUMMARY:
the efficacy and safety ofhe use of regorafenib in combination with nivolumab

DETAILED DESCRIPTION:
The present trial consists of a dose-escalation cohort to verify the tolerability of nivolumab and regorafenib when used in combination for patients with solid tumors, and to examine the clinical recommended dose(RD). The trial also consists of an expansion cohort to examine the safety and efficacy when the clinical RD is administered for several advanced solid tumors.

In the dose-escalation cohort, three patients with solid tumors will be administered 3.0 mg/kg of nivolumab once every 2 weeks and regorafenib daily for 21days, with a 1-week washout period at dose of 80 mg (level 1), 120 mg (level 2), or 160 mg (level 3). As a general rule, one cycle will last 28 days (day 1-29); however, in the event of treatment prolongation, the cycle period will be extended. The Dose Limiting Toxicity(DLT) evaluation period will be 28 days. Furthermore, for each level, three additional subjects will be added depending on the state of DLT.

In the expansion cohort, the target subject sample will consist of approximately 30 patients who will be administered 3.0 mg/kg of nivolumab once every 2 weeks, and the clinical RD of regorafenib will be determined in the dose-escalation cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who provided written informed consent to be subjects in this trial
2. Patients at least 20 years of age on the day of providing consent
3. Dose-escalation cohort: Patients with histologically or cytologically confirmed advanced or metastatic solid tumors.

   Expansion cohort: Patients with histologically or cytologically confirmed advanced or metastatic solid tumors (gastric, colorectal, or hepatocellular cancer).
4. Patients with an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1
5. Patients capable of taking oral medication
6. Patients with evaluable or measurable lesions as per RECIST version 1.1
7. Patients with adequate organ function at the time of enrollment as defined below:

   * Neutrophil count ≥1500mm3
   * Platelet count ≥10.0 × 104/mm3
   * Hemoglobin (Hb) ≥ 9 g/dL,
   * aspartate transaminase (AST), alanine transaminase (ALT) ≤100 U/L (≤100 U/L in patients with Hepatocellular carcinoma, ≤250 U/L in patients with liver metastasis)
   * Total bilirubin ≤1.5-mg /dL
   * Creatinine ≤1.5--mg /dL
   * Lipase ≤ 80 IU/L
   * Urinary protein: It satisfies one of the following (if any of the inspection criteria are satisfied, other examination may not be carried out) (i) urinary protein (test paper method) is 2+ or less (ii) Urine Protein Creatinine(UPC) ratio <3.5 (iii) 24-hour urine protein was measured, urinary protein ≦ 3500 mg
   * Prothrombin time (PT)- International normalized ratio(INR): ≤ 1.5 (≦ 3.0 in case of anticoagulant administration)
8. For women who are likely to become pregnant (including those without menstruation due to medical reasons such as chemical menopause) Note 1, we agreed to double contraceptive Note 2 for at least 5 months from consent acquisition patient to the final administration of the investigational product. Also, patients who agreed not to breast feeding for at least 5 months from acquiring consent to the final investigational drug administration.

For men, patients agreeing to double contraceptive for at least 7 months from the time of starting investigational drug administration to the final investigational drug administration.

Note 1): A woman who is likely to become pregnant is a woman who has experienced menarche and is not undergoing sterilization surgery (such as hysterectomy, bilateral salpingo ligation or bilateral oophorectomy), a woman without menopause Everything is included. The definition after menopause shall be amenorrhea continuously for 12 months or more even though there is no noteworthy reason. Women who are using oral contraceptives or mechanical contraceptive methods (such as intrauterine contraceptive devices or barrier methods) are considered to be pregnant.

Note 2): With regard to contraception, it is necessary to use two of the vasectomy or condom of a male patient or male male, the uterine tube ligation of a female patient or the other woman, a contraceptive pessary, an intrauterine contraceptive device or an oral contraceptive I need to agree to heavy contraception.

Exclusion Criteria:

1. Patients who have undergone systemic chemotherapy, radiotherapy, surgery, hormone therapy, or immunotherapy <2 weeks before enrollment. Immune checkpoint blockade as pretreatment is permitted.
2. Patients with a history of taking regorafenib.
3. Patients with hypertension that is difficult to control (systolic blood pressure ≥160 mmHg and diastolic blood pressure ≥90 mmHg) despite treatment with several hypotensive agents
4. Patients with acute coronary syndrome (including myocardial infarction and unstable angina), and with a history of coronary angioplasty or stent placement performed within 6 months before enrollment
5. Patients with a large amount of pleural effusion or ascites requiring drainage.
6. Patients with a ≥grade 3 active infection according to NCI-CTCAE version 4.03
7. Patients with symptomatic brain metastasis
8. Patients with partial or complete gastrointestinal obstruction
9. Patients with interstitial lung disease with symptoms or signs of activity
10. Patients who test positive for either anti-HIV-1 antibodies, anti-HIV-2 antibodies, hepatitis B surface antigen (HBsAg), or anti-hepatitis C virus (HCV) antibodies*

    *Patients who test positive for either anti-Hepatitis B surface(HBs) or anti- Hepatitis B core(HBc) antibodies, and those who have hepatitis B virus (HBV)-DNA measurements greater than the detection sensitivity will also be excluded.

    (However, patients with hepatocellular carcinoma in the expansion cohort will not be excluded even if they test positive for HBsAg and anti-HCV antibodies.)
11. Patients with concurrent autoimmune disease, or a history of chronic or recurrent autoimmune disease
12. Patients who require systemic corticosteroids (excluding temporary usage for tests, prophylactic administration for allergic reactions, or to alleviate swelling associated with radiotherapy) or immunosuppressants, or who have received such a therapy <14 days before enrollment in the present study
13. Patients with a history or findings of ≥grade III congestive heart failure according to the New York Heart Association functional classification
14. Patients with a seizure disorder who require pharmacotherapy
15. Patients who had grade 3 or higher bleeding during 4 weeks before enrollment
16. Patients undergoing major surgery (thoracotomy or laparotomy, etc.), laparotomy biopsy, trauma within 28 days before registration. The same day of the week before 4 weeks can be registered (However, in case of an artificial anastomosis without intestinal resection, it shall be within 14 days before registration).
17. Patients with non-healing wound, non-healing ulcer, or non-healing bone fracture.
18. Patients with a history of hypersensitivity to any of the study drugs, similar drugs, or excipients.
19. Women who are pregnant or breastfeeding, or with the potential for pregnancy.

Definition of DLT:

In principle, a DLT was any of the following Adverse Drug Reactions (ADRs) observed during Cycle 1 (28 days), which was the DLT evaluation period, and was finally determined after discussion in the coordinating committee. According to need, the opinion of the data and safety monitoring committee was to be sought.

* Hematological toxicity Grade 4 neutropenia lasting for more than 7 days. Neutrophil count of <1000/mm3 with a fever of ≥38.0°C. Grade 4 thrombocytopenia or thrombocytopenia with bleeding requiring platelet transfusion. Grade 3 thrombocytopenia with bleeding.
* Non-hematological toxicity. Grade 3 or higher non-hematological toxicity. However, non-hematological toxicities meeting any of the following criteria are classified as DLTs only when the investigator determines it impossible to continue the study even with supportive therapy.

  * Grade 3 diarrhea, nausea, vomiting, or anorexia lasting for at least 5 days.
  * Grade 3 or higher electrolyte abnormality lasting for at least 7 days.
  * Grade 3 or higher skin toxicity lasting for at least 7 days.
  * AST or ALT increased ≥5 to 8 times the upper limit of the institutional reference range that does not improve to ≤5 times the upper limit of the institutional reference range within 7 days, with T-Bil increased ≤2 times the upper limit of the institutional reference range.
  * AST or ALT increased ≥5 to 8 times the upper limit of the institutional reference range, with T-Bil increased ≥2 times the upper limit of the institutional reference range.
  * AST or ALT increased ≥8 times the upper limit of the institutional reference range.
  * T-Bil increased ≥3 times the upper limit of the institutional reference range.
  * Grade 3 or higher immune-related AEs lasting for at least 8 days even with steroid therapy.
* Overall The case in which 70% of the planned dose of regorafenib was not administered due to toxicities during the DLT evaluation period, or the case in which the specified number of nivolumab doses was not administered.

Patients evaluated for DLT:

At least 3 patients were enrolled at each dose level, and the presence or absence of a DLT was evaluated during the DLT evaluation period.

When there were patients not patient to the assessment for proceeding to the next dose level, additional patients were to be enrolled to allow the DLT evaluation specified in Section "6.1.3 Definition of DLT." Patients enrolled who met any of the following criteria were excluded from the DLT analysis set.

1. Patients in whom regorafenib was not administered for 10 days or longer during Cycle 1 for reasons other than toxicity.
2. Patients in whom no dose of nivolumab was administered during Cycle 1 for reasons other than toxicity.
3. Patients in whom adequate data for DLT evaluation were not obtained due to missing essential testing or other reasons.

Whether to include the following patients in the DLT analysis set was determined by discussion in the coordinating committee: patients who had treatment interruption with regorafenib and nivolumab during Cycle 1 for reasons other than Adverse Events (AEs) or patients who were not allowed to initiate Cycle 2 due to toxicities other than DLT.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kohei Shitara, Dr, Study Chair — National Cancer Center Hospital East
Locations (1):
- NationalCCHE, Kashiwa, Chiba, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fukuoka S, Hara H, Takahashi N, Kojima T, Kawazoe A, Asayama M, Yoshii T, Kotani D, Tamura H, Mikamoto Y, Hirano N, Wakabayashi M, Nomura S, Sato A, Kuwata T, Togashi Y, Nishikawa H, Shitara K. Regorafenib Plus Nivolumab in Patients With Advanced Gastric or Colorectal Cancer: An Open-Label, Dose-Escalation, and Dose-Expansion Phase Ib Trial (REGONIVO, EPOC1603). J Clin Oncol. 2020 Jun 20;38(18):2053-2061. doi: 10.1200/JCO.19.03296. Epub 2020 Apr 28. PMID 32343640

RESULTS

PARTICIPANT FLOW:
Recruitment Details: * 25January2018: First subject enrollment
  * 23October2018: Last subject enrollment
  * This study was conducted at second site in Japan.
  * The number of 'completers' and 'non-completers' in dose escalation cohorts will be determined by whether DLT criteria are met or not.
  * The number of cases in Expansion cohort and Dose escalation cohort who received the same dose were combined for analysis of this study.
Pre-assignment Details: *The dose escalation cohort will focus on whether the criteria for DLT evaluation were met in the first cycle, i.e., safety in the first cycle, while the final analysis of the expansion cohort will focus on clinical efficacy and safety in all cycles.
  **The planned number of cases in this clinical trial was 9 to 18 in the dose escalation cohort and approximately 30 in the expansion cohort, but the actual number was 14 in the dose escalation cohort and 36 in the expansion cohort.
Groups:
- Regorafenib 80mg/Day: Regorafenib: Oral administration at a dose of 80 mg/day for 21 consecutive days, with a 1-week washout period.
  Nivolumab at a dose of 3.0 mg/kg was administered once every 2 weeks. With 1 cycle being 28 days, the treatment was repeated until any of the discontinuation criteria was met.
  After starting the trial, three cases are enrolled for each dose level, and temporary case registration is suspended until safety evaluation of the first course is completed in all cases. If tolerability at level 1 is confirmed, confirm the tolerability at level 2.
  In addition, if there are patients who are not eligible for level transition, additional patients will be enrolled so that DLT evaluation can be performed.
  For the dose-escalation method, see Section "Outcome Measure Description" in " 1. Primary Outcome".
- Regorafenib 120mg/Day: Regorafenib: Oral administration at a dose of 120 mg/day for 21 consecutive days, with a 1-week washout period.
  Nivolumab at a dose of 3.0 mg/kg was administered once every 2 weeks. With 1 cycle being 28 days, the treatment was repeated until any of the discontinuation criteria was met.
  After starting the trial, three cases are enrolled for each dose level, and temporary case registration is suspended until safety evaluation of the first course is completed in all cases. If tolerability at level 2 is confirmed, confirm the tolerability at level 3.
  In addition, if there are patients who are not eligible for level transition, additional patients will be enrolled so that DLT evaluation can be performed.
  For the dose-escalation method, see Section "Outcome Measure Description" in " 1. Primary Outcome".
- Regorafenib 160mg/Day: Regorafenib was administered once daily at a dose of 160 mg/day for 21 consecutive days, followed by a 1-week rest period.
  Nivolumab at a dose of 3.0 mg/kg was administered once every 2 weeks. With 1 cycle being 28 days, the treatment was repeated until any of the discontinuation criteria was met.
  After starting the trial, three cases are enrolled for each dose level, and temporary case registration is suspended until safety evaluation of the first course is completed in all cases. If tolerability at level 3 is confirmed, set the doses at level 3 as Recommended Dose (RD).
  For the dose-escalation method, see Section "Outcome Measure Description" in" 1. Primary Outcome".
Period: Dose Escalation Cohort
Arm/Group | Regorafenib 80mg/Day | Regorafenib 120mg/Day | Regorafenib 160mg/Day
Started | 4 | 7 | 3
Completed | 3 | 6 | 3
Not Completed | 1 | 1 | 0
Not completed — DLT assesment cancellation** | 1 | 1 | 0
Period: Expansion Cohort(Final Analysis)
Arm/Group | Regorafenib 80mg/Day | Regorafenib 120mg/Day | Regorafenib 160mg/Day
Started | 22 | 25 | 3
Completed | 0 | 0 | 0
Not Completed | 22 | 25 | 3
Not completed — Completion of 54 doses of Nivolumab | 4 | 2 | 1
Not completed — Progression of primary disease | 17 | 22 | 1
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Death | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: * This clinical trial was divided into a dose-escalation cohort to determine RD based on the number of DLTs, and an expansion cohort to evaluate the efficacy and safety of this regimen based on RD. Patient Background data were combined from both cohorts and presented as final analysis data.
  * Stastical analyses by tumor were not performed, because this clinical trial did not use a randomized design.
Groups:
- Final Analysis: Regorafenib 80mg/Day: Regorafenib: One course will last 28 days. Oral administration at a dose of Regorafenib 80mg/day for 21 consecutive days, with a 1-week washout period.
  Nivolumab at a dose of 3.0 mg/kg was administered once every 2 weeks.
  With 1 cycle being 28 days, the treatment was repeated until any of the discontinuation criteria was met.
  Follow the instructions in this clinical protocol to suspend and resume administration.
- Final Analysis: Regorafenib 120mg/Day: Regorafenib: One course will last 28 days. Oral administration at a dose of 120mg/day for 21 consecutive days, with a 1-week washout period.
  Nivolumab at a dose of 3.0 mg/kg was administered once every 2 weeks.
  With 1 cycle being 28 days, the treatment was repeated until any of the discontinuation criteria was met.
  Follow the instructions in this clinical protocol to suspend and resume administration.
- Final Analysis: Regorafenib 160mg/Day: Regorafenib: One course will last 28 days. Oral administration at a dose of 160mg/day for 21 consecutive days, with a 1-week washout period.
  Nivolumab at a dose of 3.0 mg/kg was administered once every 2 weeks.
  With 1 cycle being 28 days, the treatment was repeated until any of the discontinuation criteria was met.
  Follow the instructions in this clinical protocol to suspend and resume administration.
- Total: Total of all reporting groups
Arm/Group | Final Analysis: Regorafenib 80mg/Day | Final Analysis: Regorafenib 120mg/Day | Final Analysis: Regorafenib 160mg/Day | Total
Number analyzed (Participants) | 22 | 25 | 3 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 17 | 2 | 31
  >=65 years | 10 | 8 | 1 | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 1 | 10
  Male | 17 | 21 | 2 | 40
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 22 | 25 | 3 | 50

OUTCOME MEASURES:

1. Primary Outcome: The Number of Dose Limiting Toxicity (DLT) for RD Determination
Description: The procedure for DLT assessment was as follows:
  1. When DLT is observed in 1 out of 3 cases, 3 additional cases are added to the administration level.
  2. When DLT is observed in more than 2 of 3 cases, it is judged that the administration level exceeds Maximum Tolerated Dose (MTD).
  3. If the number of DLT is 1 case or less in 6 cases, shift to the next level.
  4. If MTD is exceeded, shift to the next lower level. At the relevant dose, if only 3 people are evaluating DLT, add 3 cases. When the number of DLT is 1 or less out of 6, the dose is defined as MTD and RD. If it is judged that Level 1 exceeds the MTD, review the dose or consider stopping the trial.
  5. MTD should be the highest dose level of DLT expression less than 1 in 6 cases. - After the RD was determined and the patient moved to the expansion cohort, G3 skin toxicity occurred, so based on the recommendation of the Data and Safety Monitoring Committee, the RD was reduced by one level and the trial was resumed.
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Dose Escalation Cohort Regorafenib 80mg: Regorafenib: One course will last 28 days. Oral administration at a dose of 80 mg/day for 21 consecutive days, with a 1-week washout period.
  Nivolumab at a dose of 3.0 mg/kg was administered once every 2 weeks.
  With 1 cycle being 28 days, the treatment was repeated until any of the discontinuation criteria was met.
  Register 3 cases first at each dose level, and temporarily suspend case registration until the safety assessment of the first course of all cases is completed. If no DLT is observed in 3 cases, proceed to the next dose level. If DLT is not observed in 3 cases of level 3, add 3 more cases to this level (total 6 cases).
  In addition, if there are patients who are not eligible for level transition, additional patients will be enrolled so that DLT evaluation can be performed.
- Dose Escalation Cohort Regorafenib 120mg: Regorafenib: One course will last 28 days. Oral administration at a dose of 120 mg/day for 21 consecutive days, with a 1-week washout period.
  Nivolumab at a dose of 3.0 mg/kg was administered once every 2 weeks.
  With 1 cycle being 28 days, the treatment was repeated until any of the discontinuation criteria was met.
  At least 3 patients were enrolled at each dose level, and the presence or absence of a DLT was evaluated during the DLT evaluation period.
  When there were patients not patient to the assessment for proceeding to the next dose level, additional patients were to be enrolled to allow the DLT evaluation. If there are cases in which evaluation of DLT can not be performed properly, such as being canceled due to reasons other than safety during the course of the first course, the necessary number of cases is appropriately added to the administration level.
  In addition, if there are patients who are not eligible for level transition, additional patients will be enrolled so that DLT evaluation can be performed.
- Dose Escalation Cohort Regorafenib 160mg: Regorafenib: One course will last 28 days. Oral administration at a dose of 160 mg/day for 21 consecutive days, with a 1-week washout period.
  Nivolumab at a dose of 3.0 mg/kg was administered once every 2 weeks.
  With 1 cycle being 28 days, the treatment was repeated until any of the discontinuation criteria was met.
  If it is judged that MTD is exceeded, 6 cases of DLT evaluation are already carried out at the level one level below and if the DLT is 1 case or less of 6 cases, the dose is taken as MTD and RD. At the relevant dose, if only 3 people are evaluating DLT, add 3 cases (total 6 cases). When the number of DLT is 1 or less out of 6, the dose is defined as MTD and RD.
- Expansion Cohort : Regorafenib 120mg: Regorafenib: One course will last 28 days. Oral administration for 21 consecutive days, with a 1-week washout period. As for the expansion cohort, implemented using the RD estimated in the dose-escalation cohort.
  Nivolumab: One course will last 28 days. Given once every 2 weeks at a dose of 3.0 mg/kg.
  After moving to the expansion cohort, G3 skin-related toxicity occurred, and RD was reduced by one level based on the recommendation of the Data and Safety Monitoring Committee as specified in this clinical protocol.
Arm/Group | Dose Escalation Cohort Regorafenib 80mg | Dose Escalation Cohort Regorafenib 120mg | Dose Escalation Cohort Regorafenib 160mg | Expansion Cohort : Regorafenib 120mg
Number analyzed (Participants) | 3 | 6 | 3 | 18
Participants | 0 | 0 | 3 | 5

2. Secondary Outcome: Objective Response Rate (ORR)
Description: *Objective Response Rate is defined as the proportion of patients whose best overall response, as per the Response Evaluation Criteria in Solid Tumors (RECIST) guideline version 1.1 and immune-related RECIST (irRECIST), is either Complete Response (CR) or Partial Response (PR).
Time Frame: 2year
Population: The primary objective of this study was to evaluate the RD on the basis of the safety of the combination of nivolumab and regorafenib, and the clinical trial was intended to evaluate the efficacy of this therapy secondarily. Therefore, dose-specific efficacy analyses were not preplanned or considered to evaluate this outcome measure. Ultimately, the trial was intended to provide an overall efficacy in this study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Final Analysis: Regorafenib was administered once daily for 21 consecutive days, followed by a 1-week treatment interruption.
  Nivolumab at a dose of 3.0 mg/kg was administered once every 2 weeks.
  With 1 cycle being 28 days, the treatment was repeated until any of the discontinuation criteria was met.
  Expansion cohort: Implemented using the RD estimated in Dose-escalation cohort. In Expansion cohort, skin toxicity occurred, so based on the recommendation of Data and Safety Monitoring Committee, the RD was reduced by one level and the trial was resumed.
Arm/Group | Final Analysis
Number analyzed (Participants) | 50
percentage of participants | 42.0 [28.2 to 56.8]

3. Secondary Outcome: Progression-Free Survival(PFS)
Description: *PFS is defined as the time from the enrollment date to either the date when disease progression is determined or the date of death from any cause, whichever came earlier.
  The data were compiled according to the analysis plan outlined in the protocol. No analysis was conducted to determine efficacy by cancer type or dose level.
Time Frame: 6 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Final Analysis
Number analyzed (Participants) | 50
months | 6.3 [3.9 to 10.4]

4. Secondary Outcome: Overall Survival(OS)
Description: *OS is defined as the period from the date of enrollment to the date of death from any cause.
  Surviving patients are censored on the last confirmation date of survival (confirmation of survival by telephone is permitted; the fact that survival is confirmed is to be recorded in the medical record, etc.).
  Patients lost to follow-up are censored on the last date on which their survival is confirmed before being lost to follow-up.
  The data were compiled according to the analysis plan outlined in the protocol. No analysis was conducted to determine efficacy by cancer type or dose level.
Time Frame: 2year
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: median of months
Arm/Group | Final Analysis
Number analyzed (Participants) | 50
median of months | 14.4 [9.8 to 21.7]

5. Secondary Outcome: Disease Control Rate(DCR)
Description: *DCR is defined as the proportion of patients whose best overall response assessed based on the RECIST guideline version 1.1 and irRECIST is any of CR, PR, or Stable Disease (SD).
  The data were compiled according to the analysis plan outlined in the protocol. No analysis was conducted to determine efficacy by cancer type or dose level.
Time Frame: 2year
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Final Analysis
Number analyzed (Participants) | 50
percentage of participants | 86.0 [73.3 to 94.2]

6. Secondary Outcome: Adverse-Events
Description: * The occurrences rate of each AE of the worst grade occurring in this study was evaluated based on the Common Terminology Criteria for Adverse Events (CTCAE) v4.03 throughout the entire cycles will be calculated. Additionally, this study included a special note regarding abnormal laboratory values. If clinical signs and symptoms observed in this study were induced, the diagnosis and associated data were collected based on whether or not they were due to abnormal laboratory values. Therefore, for example, results of grading regarding liver dysfunction may differ between non-hematologic toxicity and laboratory values.
  * Adverse-Events occurrences means "prevalence proportion" of any undesirable occurrence based on investigator's medical decision in this study.
Time Frame: 2 year
Population: This protocol specifies that secondary endpoint were not analysed separately for colorectal cancer and gastric cancer, and cases both the dose escalation cohort and the expansion cohort were included.
Measure: Count of Participants; unit: Participants
Groups:
- Final Analysis: Regorafenib 80mg: Regorafenib: One course will last 28 days. Oral administration at a dose of 80 mg/day for 21 consecutive days, with a 1-week washout period.
  Nivolumab at a dose of 3.0 mg/kg was administered once every 2 weeks.
  With 1 cycle being 28 days, the treatment was repeated until any of the discontinuation criteria was met.
- Final Analysis: Regorafenib 120mg: Regorafenib: One course will last 28 days. Oral administration at a dose of 120mg/day for 21 consecutive days, with a 1-week washout period.
  Nivolumab at a dose of 3.0 mg/kg was administered once every 2 weeks.
  With 1 cycle being 28 days, the treatment was repeated until any of the discontinuation criteria was met.
  Given once every 2 weeks at a dose of 3.0 mg/kg.
- Final Analysis: Regorafenib 160mg: Regorafenib: One course will last 28 days. Oral administration at a dose of 160 mg/day for 21 consecutive days, with a 1-week washout period.
  Nivolumab at a dose of 3.0 mg/kg was administered once every 2 weeks.
  With 1 cycle being 28 days, the treatment was repeated until any of the discontinuation criteria was met.
Arm/Group | Final Analysis: Regorafenib 80mg | Final Analysis: Regorafenib 120mg | Final Analysis: Regorafenib 160mg
Number analyzed (Participants) | 22 | 25 | 3
Participants | 22 | 25 | 3

ADVERSE EVENTS:
Time Frame: 2 year, 2months
Description: *Adverse events were not analyzed separately for colorectal cancer and gastric cancer.
Groups:
- Final Analysis: Regorafenib 80mg/Day: Regorafenib: One course will last 28 days. Oral administration at a dose of 80 mg/day for 21 consecutive days, with a 1-week rest period.
  Nivolumab: One course will last 28 days. Given once every 2 weeks at a dose of 3.0 mg/kg.
  With 1 cycle being 28 days, the treatment was repeated until any of the discontinuation criteria was met.
- Final Analysis: Regorafenib 120mg/Day: Regorafenib: One course will last 28 days. Oral administration at a dose of 120mg/day for 21 consecutive days, with a 1-week rest period.
  Nivolumab: One course will last 28 days. Given once every 2 weeks at a dose of 3.0 mg/kg.
  With 1 cycle being 28 days, the treatment was repeated until any of the discontinuation criteria was met.
- Final Analysis: Regorafenib 160mg: Regorafenib: One course will last 28 days. Oral administration at a dose of 160 mg/day for 21 consecutive days, with a 1-week rest period.
  Nivolumab: One course will last 28 days. Given once every 2 weeks at a dose of 3.0 mg/kg.
  With 1 cycle being 28 days, the treatment was repeated until any of the discontinuation criteria was met.
Arm/Group | Final Analysis: Regorafenib 80mg/Day | Final Analysis: Regorafenib 120mg/Day | Final Analysis: Regorafenib 160mg
All-Cause Mortality (participants affected / at risk) | 0/22 | 1/25 | 0/3
Serious Adverse Events (participants affected / at risk) | 4/22 | 5/25 | 2/3
Other Adverse Events (participants affected / at risk) | 22/22 | 25/25 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Final Analysis: Regorafenib 80mg/Day (N=22) | Final Analysis: Regorafenib 120mg/Day (N=25) | Final Analysis: Regorafenib 160mg (N=3)
rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
large intestine perforation (Gastrointestinal disorders) | 1 | 0 | 1
death (General disorders) | 0 | 1 | 0
erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
diarrhea (Gastrointestinal disorders) | 0 | 1 | 0
fever (General disorders) | 0 | 1 | 0
abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
hypopituitarism (Endocrine disorders) | 1 | 0 | 0
Guillain-Barre syndrome (Nervous system disorders) | 1 | 0 | 0
interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
malaise (General disorders) | 1 | 0 | 0
hyperglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Final Analysis: Regorafenib 80mg/Day (N=22) | Final Analysis: Regorafenib 120mg/Day (N=25) | Final Analysis: Regorafenib 160mg (N=3)
palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 13 | 20 | 2
hypertension (Vascular disorders) | 11 | 14 | 0
malaise (General disorders) | 11 | 10 | 2
fever (General disorders) | 10 | 10 | 1
proteinuria (Renal and urinary disorders) | 6 | 9 | 2
decreased appetite (Metabolism and nutrition disorders) | 6 | 7 | 1
maculo-papular rash (Skin and subcutaneous tissue disorders) | 3 | 8 | 1
stomatitis (Gastrointestinal disorders) | 4 | 6 | 2
diarrhea (Gastrointestinal disorders) | 6 | 4 | 2
Liver disorders (Hepatobiliary disorders) | 4 | 6 | 0
hypothyroidism (Endocrine disorders) | 5 | 2 | 0
platelet count decreased (Investigations) | 1 | 5 | 1
asparate aminotaransferase increased (Investigations) | 1 | 2 | 0
dysphonia (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 0
hyperthyroidism (Endocrine disorders) | 4 | 2 | 0
weight decreased (Investigations) | 5 | 2 | 1
pneumonia (Infections and infestations) | 2 | 1 | 0
neutrophil count decreased (Investigations) | 1 | 2 | 0
nasopharygititis (Infections and infestations) | 4 | 3 | 0
rash (Skin and subcutaneous tissue disorders) | 7 | 4 | 1
back pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1 | 0
arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 3 | 0
anemia (Blood and lymphatic system disorders) | 4 | 1 | 0
constipation (Gastrointestinal disorders) | 3 | 1 | 0
fatigue (General disorders) | 2 | 2 | 0
alanine aminotransferase increased (Investigations) | 1 | 2 | 0
blood bilirubin increased (Investigations) | 0 | 2 | 1
blood creatinine phosphokinase increased (Investigations) | 1 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-20): https://cdn.clinicaltrials.gov/large-docs/71/NCT03406871/Prot_SAP_000.pdf